CLINICAL TRIAL: NCT06343584
Title: Are Personal Smartphones Hurting Work-Life Balance for Nurse Managers?
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 023.NUR.2021.M
Record Dates: First submitted 2022-04-27; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2022-04

CONDITIONS: Burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Must hold the title of Nurse Manager or Interim Nurse Manager at Methodist Mansfield Medical Center. Upon receipt of informed consent, participants will be divided into two groups.
  Group 1 will receive a list of suggested tools used to decrease the amount of smartphone interruptions after business hours
  Interventions: Other: Study will conducted over a six-month period using a quasi-experimental Pre-test/Post-test design using Stamm's (2009) ProQOL Scale.
- Group 2: Must hold the title of Nurse Manager or Interim Nurse Manager at Methodist Mansfield Medical Center. Upon receipt of informed consent, participants will be divided into two groups.
  Group 2 will receive a work-issued smartphone with instructions for use (Appendix C).
  Interventions: Other: Study will conducted over a six-month period using a quasi-experimental Pre-test/Post-test design using Stamm's (2009) ProQOL Scale.

INTERVENTIONS:
Other: Study will conducted over a six-month period using a quasi-experimental Pre-test/Post-test design using Stamm's (2009) ProQOL Scale. — Group 1 will receive a list of suggested tools used to decrease the amount of smartphone interruptions after business hours (Appendix B) and Group 2 will receive a work-issued smartphone with instructions for use (Appendix C). Both groups will use a pre-post test format designed to compare the outcomes between the two groups. Post-study analysis will compare pre- and post-tests within each group and will compare Group 1 and Group 2 post-intervention outcomes.

SUMMARY:
For leadership positions with only a handful of staff under their direct chain of command, this may not be all-consuming and detrimental to work-life balance. But for NMs with upwards of 100 direct reports, this can make for a never-ending stream of contact points. This study will implement several communication and behavioral strategies to determine how using provided smartphone tools impact work-life balance and professional burnout.

DETAILED DESCRIPTION:
The study will be conducted over a six-month period using a quasi-experimental Pre-test/Post-test design using Stamm's (2009) ProQOL Scale. This study is being done as a pilot study with a small sample size. NMs will be recruited as volunteers for participation in the study with an anticipated six-month time commitment. Upon receipt of informed consent, participants will be divided into two groups. Group 1 will receive a list of suggested tools used to decrease the amount of smartphone interruptions after business hours (Appendix B) and Group 2 will receive a work-issued smartphone with instructions for use (Appendix C). Both groups will use a pre-post test format designed to compare the outcomes between the two groups. Post-study analysis will compare pre- and post-tests within each group and will compare Group 1 and Group 2 post-intervention outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participant must hold the title of Nurse Manager or Interim Nurse Manager at Methodist Mansfield Medical Center
* Participant must have greater than 50 direct reports

Exclusion Criteria:

* Participant expects to separate employment with Methodist Health System prior to the conclusion of the study
* Participant does not use their personal smartphone to communicate with direct reports

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Participant must hold the title of Nurse Manager or Interim Nurse Manager at Methodist Mansfield Medical Center
  * Participant must have greater than 50 direct reports
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
• Impact of smartphone tool utilization will be measured using a pre-study survey and post-study survey using the Professional Quality of Life (ProQOL) Scale (Stamm, 2009). | 6 months
  • Impact of smartphone tool utilization will be measured using a pre-study survey and post-study survey using the Professional Quality of Life (ProQOL) Scale (Stamm, 2009).

SECONDARY OUTCOMES:
• Participants in Group 1 will self-report on the post-study survey (Appendix D1) the number of tools implemented during the study duration. | 6 months
  • Participants in Group 1 will self-report on the post-study survey (Appendix D1) the number of tools implemented during the study duration.
• Participants in Group 1 will self-report on the post-study survey (Appendix D1) the frequency of tool utilization during the study duration using a Likert scale. | 6 months
  • Participants in Group 1 will self-report on the post-study survey (Appendix D1) the frequency of tool utilization during the study duration using a Likert scale.
• Participants in Group 2 will self-report on the post-study survey (Appendix D2) using the ProQOL Scale. | 6 months
  • Participants in Group 2 will self-report on the post-study survey (Appendix D2) using the ProQOL Scale.
• Responses to the post-study survey from participants in Group 2 will be compared to participants in Group 1 to determine if utilizing a separate work smartphone during business hours has a greater improvement on work-life balance and burnout. | 6 months
  • Responses to the post-study survey from participants in Group 2 will be compared to participants in Group 1 to determine if utilizing a separate work smartphone during business hours has a greater improvement on work-life balance and burnout.

CONTACTS AND LOCATIONS:
Overall Officials: Brooks Williams, DNP, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Mansfield Medical Center, Mansfield, Texas, United States